CLINICAL TRIAL: NCT03242694
Title: Left Atrial Function Analysis With Multimodal Techniques for Patients With Persistent Atrial Fibrillation Undergoing Pulmonary Vein Isolation
Brief Title: Left Atrial Function Analysis for Patients With Persistent Atrial Fibrillation Undergoing Pulmonary Vein Isolation
Acronym: LAMPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: LAMPP 1.0
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Persistent Atrial Fibrillation; Catheter Ablation
Keywords: persistent atrial fibrillation; pulmonary vein isolation; catheter ablation; left atrial function; left atrial pressure; voltage map; strain; scar; success; biomarker
MeSH Terms: conditions — Atrial Fibrillation; Sprains and Strains; Cicatrix | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- persistent atrial fibrillation: invasive LA pressure monitoring, LA voltage map creation, LA strain evaluation by transthoracal echocardiography, LA scar-mapping by cardiac MRI, defining biomarkers from blood samples during atrial fibrillation and after pulmonary vein isolation in sinus rhythm
  Interventions: Diagnostic Test: LA pressure, voltage map, strain, scar-map, blood sampling; Procedure: pulmonary vein isolation

INTERVENTIONS:
Diagnostic Test: LA pressure, voltage map, strain, scar-map, blood sampling — invasive LA pressure monitoring, LA voltage map creation, LA strain evaluation by transthoracal echocardiography, LA scar-mapping by cardiac MRI, defining biomarkers from blood samples during atrial fibrillation and after pulmonary vein isolation in sinus rhythm
Procedure: pulmonary vein isolation — pulmonary vein isolation without creating additional ablation lesions

SUMMARY:
This prospective observational study is designed to describe the factors determining the success of pulmonary vein isolation (PVI) for patients with persistent atrial fibrillation (AF). These factors - described as left atrial (LA) function - are simultaneously studied by multi-modal techniques in patients undergoing radiofrequency ablation. The simultaneous measurements are conducted before the PVI in AF and after the sinus rhythm converted due to PVI. These measurements include invasive LA pressure monitoring, LA voltage map creation, LA strain evaluation by transthoracal echocardiography, LA scar-mapping by cardiac MRI, defining biomarkers from blood samples. During the one year follow-up period rhythm monitoring is conducted by regular Holter-monitoring. Our aim is to define the predictive values of the above mentioned factors and to create a new score system for predicting PVI success in persistent AF population.

ELIGIBILITY:
Inclusion Criteria:

* documented, symptomatic persistent atrial fibrillation (AF)
* catheter ablation is indicated
* aged 18-75 years
* signed Patient Informed Consent Form
* able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* secondary AF
* paroxysmal, long-standing persistent or permanent AF
* ejection fraction < 30%
* GFR <30 ml/min/1.73m2
* unstable angina pectoris or myocardial infarction within the past 2 months
* severe heart failure (NYHA IV)
* severe COPD (GOLD III-IV)
* previous left atrial catheter ablation
* previous transthoracic cardiac surgery
* implanted cardiac device (pacemaker, ICD, CRT, VAD)
* awaiting cardiac transplantation or other cardiac surgery within the next 12 months
* any contraindication for pulmonary vein isolation, MRI or anticoagulation
* coagulopathy
* active malignancy, left atrial myxoma
* autoimmune disorder, chronic inflammatory disease
* acute illness, active systemic infection, sepsis
* women who are pregnant, breast feeding, or planning to become pregnant in the next 12 months
* aged under 18 years or above 75 years
* enrollment in other studies, which exclude participation in other studies
* patient not willing or not able to sign the informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent atrial fibrillation referred for pulmonary vein isolation at Heart and Vascular Center of Semmelweis University, Budapest, Hungary.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
one-year success of pulmonary vein isolation | 3-12 months after the first pulmonary vein isolation
  one-year success without recurrent atrial fibrillation or atrial tachycardia without antiarrhythmic drugs after the three-month blanking period of pulmonary vein isolation

SECONDARY OUTCOMES:
acute unsuccessful pulmonary vein isolation | within 5 minutes after the last application is performed at the ablation procedure
  operator is unable to disconnect pulmonary veins from the left atrium
usage of antiarrhythmic drugs after the three-month blanking period | 3-12 months after the first pulmonary vein isolation
  antiarrhythmic drugs: sotalol, amiodarone, propafenon
reablation | 3-12 months after the first pulmonary vein isolation
  repeated left atrial ablation is performed due to atrial fibrillation or left atrial tachycardia recurrence
major complications of pulmonary vein isolation | through 1 year follow-up after the first pulmonary vein isolation
  major complications: requiring surgical intervention or causing prolonged hospitalisation
MACE | through 1 year follow-up after the first pulmonary vein isolation
  major adverse cardiac events
death | through 1 year follow-up after the first pulmonary vein isolation

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Geller, MD PhD, Principal Investigator — Heart and Vascular Center of Semmelweis University; Bela Merkely, MD PhD DSc, Study Director — Heart and Vascular Center of Semmelweis University
Locations (1):
- Heart and Vascular Center of Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No